CLINICAL TRIAL: NCT03127865
Title: Evaluation of Electrical Velocimetry for Assessment of Extra-vascular Lung Water in Pre-eclamptic Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Lecturer of anesthesia and critical care medicine, Cairo University
Other Study IDs: N-28-2017
Record Dates: First submitted 2017-04-12; First posted 2017-04-25 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to compare the sensitivity and the specificity of electrical cardiometry to the lung ultrasound in measuring thoracic lung water in pregnant females with pre-eclampsia. If electrical cardiometry is validated against ultrasound, it will be easy to use with numerical number that will not require advanced experience as with the ultrasound.

DETAILED DESCRIPTION:
Pre-eclampsia is accompanied with increased risk of serious complications such as pulmonary edema, cerebrovascular accidents, coagulopathy, and hemorrhage.

Pre-eclampsia is responsible for 46.6% of the etiology of acute pulmonary edema in pregnant women.

Fluid management in pre-eclamptic patients is challenging. Hypovolemia exacerbates organ failure, whereas volume overload results in pulmonary edema. Thus, using different methods for evaluation of volume status of the patients would improve patient management. Lung ultrasound has been developed as an accurate non-invasive method for assessment of extra-vascular lung water; However, ultrasound needs skilled operator. Electrical velocimetry (cardiometry) is a newer technology for assessment of total thoracic fluid content (TFC); however, it has not been validated in pre-eclamptic patients.

In this study the investigators will validate the accuracy of cardiometry in evaluation of lung water using the lung ultrasound as a gold standard. Both methods will be evaluated for prediction of the need of diuretic therapy and the need for post-operative oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* pre-eclamptic
* In first stage of labor

Exclusion Criteria:

* Eclampsia.
* Second, third and fourth stages of labor on admission.
* Patients with severe cardiac and/or pulmonary disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-eclamptic patients scheduled for normal vaginal delivery or casearen section
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
total thoracic fluid content | after 30 minutes from patient admission to the obstetric casuality
  total fluid content measured by electrical velocimetry device (cardiometry)

SECONDARY OUTCOMES:
The need of diuretics | during the period starting from admission till one day after delivery
  The presence of lung congestion manifested by respiratory distress (dyspnea, tachypnea, and decreased oxygen saturation below 90%) needing intravenous diuretics
extra-vascular lung water | after 30 minutes from patient admission to the obstetric casuality
  extra-vascular lung water measured by ultrasound (lung ultrasound score)
lung congestion | during the period starting from admission till one day after delivery
  the presence of lung congestion manifested by audible crepitations by chest auscultation
serum albumin | after 30 minutes from patient admission to the obstetric casuality
  the level of albumin in blood (measured by g/ liter
arterial blood pressure | after 30 minutes from patient admission to the obstetric casuality
  arterial blood pressure measured in mmHg
heart rate | after 30 minutes from patient admission to the obstetric casuality
  the number of heart beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Chair — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No